CLINICAL TRIAL: NCT03951324
Title: Volumetric Laser Endomicroscopy's (VLE) Diagnostic Accuracy Validation Study: Impact on Clinical Management Study
Acronym: VLE-IOV
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Innovative Digestive Health Education and Research Inc (Other)
Collaborators: NinePoint Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 2565207-44318141
Record Dates: First submitted 2019-05-13; First posted 2019-05-15 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Biliary Stricture; Pancreas Cancer; Cholangiocarcinoma; Bile Duct Cancer; Bile Duct Neoplasms Malignant; Bile Duct Neoplasms; Bile Duct Lesions; Bile Duct Obstruction; Bile Duct Diseases; Bile Duct Obstruction, Extrahepatic; Bile Duct Stenosi; Bile Duct Adenoma; Pancreatic Duct Stricture; Pancreatic Duct Stenosis; Pancreatic Duct Obstruction; Pancreatic Ductal Adenocarcinoma; Primary Sclerosing Cholangitis
Keywords: bile duct stricture; bile duct neoplasm; bile duct obstruction; bile duct lesion; cholangiocarcinoma; pancreatic duct stricture; pancreatic duct obstruction; pancreatic cancer; primary sclerosing cholangitis
MeSH Terms: conditions — Pancreatic Neoplasms; Cholangiocarcinoma; Bile Duct Neoplasms; Cholestasis; Bile Duct Diseases; Cholestasis, Extrahepatic; Adenoma, Bile Duct; Cholangitis, Sclerosing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Expert Endoscopists: Experienced Endoscopists with significant user experience with Volumetric Laser Endomicroscopy for bile duct/pancreatic duct strictures
  Interventions: Other: Interobserver agreement or Interrater agreement
- None-Expert Endoscopists: Experienced Endoscopists with non-significant or beignner user experience with Volumetric Laser Endomicroscopy for bile duct/pancreatic duct strictures
  Interventions: Other: Interobserver agreement or Interrater agreement

INTERVENTIONS:
Other: Interobserver agreement or Interrater agreement — Interobserver agreement or Interrater agreement using 9 visual criteria for diagnosing VLE clips that feature indeterminate biliary or pancreatic duct strictures

SUMMARY:
The purpose of this study is to assess the interobserver agreement (IOV) for pancreatico-biliary Volumetric Laser Endomicroscopy (VLE) de-identified clips using the new VLE criteria.

This is an Interobserver study to validate VLE criteria for indeterminate biliary and pancreatic duct strictures and evaluate impact on clinical management.

DETAILED DESCRIPTION:
Objective: Validate diagnostic impact of VLE diagnostic accuracy on clinical management

Primary Objectives:

1. Interobserver study for criteria validation and accuracy, Positive predictive value (PPV) and Negative predictive value (NPV), sensitivity and specificity.
2. Evaluation of VLE diagnostics on clinical management (increased accuracy/faster detection)
3. Determination of learning curve to standardize credentialing for endoscopists to use and interpret VLE imaging for biliary/pancreatic treatment management.

B. Hypotheses / Research Question(s) The new VLE criteria for biliary and pancreatic duct strictures increase accuracy, thus leading to substantial impact on clinical management (Screening and Treatment)

Study Design (2 phase):

* Phase 1: Primary Objective 1 and 2 part of the study will be completed.
* Phase 2: Primary Objective 3 of the study will be conducted within 1 month.

Study Timeline: 3 months post WIRB approval. Sample size: 40 VLE Clips of at least 20 seconds featuring one or more the VLE criteria. All clips will have confirmed diagnosis for accuracy analysis. All clips will be de-identified. All clips will be removed from RedCAP and other secure cloud storage upon completion of study.

Clips will be supplied by NinePoint Medical, the company behind VLE OCT. All VLE clips will be from a dataset of clips collected from adults > 18 and who underwent Endoscopic retrograde cholangiopancreatography (ERCP) with indeterminate biliary stricture indications. The clips are chosen based on the quality of the clips, duration, final diagnosis and presence of either benign or malignant criteria.

Investigators: Up to 30 Expert and non-expert endoscopists currently using VLE

ELIGIBILITY:
Inclusion Criteria:

VLE clips featuring indeterminate biliary or pancreatic duct stricture with confirmed diagnosis on pathology -

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: VLE clips featuring indeterminate biliary or pancreatic duct stricture with confirmed diagnosis on pathology.
  Endoscopists who use VLE to diagnose indeterminate biliary or pancreatic duct strictures.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Interobserver agreement and diagnostic accuracy | 2 months
  Interobserver study for criteria validation and accuracy, PPV and NPV, sensitivity and specificity
Frequency and type of criteria visually identified on malignant VLE clips | 2 months
  Correlation analysis of any of the 9 visual criteria with malignancy diagnosis as determined by endoscopist

SECONDARY OUTCOMES:
Number of procedures needed to view and conduct to use VLE for diagnostic confirmation | 2 months
  Learning curve using CUSUM analysis to standardize credentialing for endoscopists to use and interpret VLE imaging for biliary/pancreatic treatment management proficiently.

CONTACTS AND LOCATIONS:
Overall Officials: Michel Kahaleh, MD, Principal Investigator — Innovative Digestive Health Education and Research Inc
Locations (1):
- Innovative Digestive Health Education & Research Inc, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided